CLINICAL TRIAL: NCT06903858
Title: Neoadjuvant Toripalimab Plus Celecoxib in Mismatch-repair Deficient or Microsatellite Instability-high Locally Advanced Colorectal Cancer (PICC-3): a Multicenter, Single-arm, Phase 2 Trial
Brief Title: Neoadjuvant Toripalimab Plus Celecoxib for dMMR/MSI-H Locally Advanced Colorectal Cancer
Acronym: PICC-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG-C08
Record Dates: First submitted 2025-03-28; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC); PD-1 Inhibitor; Neoadjuvant Immunotherapy; Celecoxib; Watch &Amp; Wait
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, Single-arm, Phase II
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Toripalimab plus Celecoxib (Experimental): Neoadjuvant Treatment Phase Toripalimab is administered via intravenous infusion at 3 mg/kg over 30 minutes (initial infusion time is 60 minutes), once every two weeks, for a total of 12 doses before surgery. Celecoxib is taken orally at 200 mg per dose, twice daily, for a duration of 6 months.
  Assessment After Neoadjuvant Treatment
  1. Patients achieving clinical complete response (cCR) based on radiographic imaging (CT/MRI of chest, abdomen, pelvis, and rectal MRI), endoscopy, and digital rectal examination (if applicable) are recommended to adopt a watch-and-wait strategy.
  2. Patients who do not achieve cCR based on radiographic imaging (CT/MRI of chest, abdomen, pelvis, and rectal MRI), endoscopy, and digital rectal examination (if applicable) are recommended to undergo curative resection of colorectal cancer.
  Interventions: Drug: Toripalimab combined with celecoxib; Procedure: Curative resection of colorectal cancer; Other: Watch-and-wait strategy

INTERVENTIONS:
Drug: Toripalimab combined with celecoxib — Toripalimab is administered via intravenous infusion at 3 mg/kg over 30 minutes (initial infusion time is 60 minutes), once every two weeks, for a total of 12 doses before surgery. Celecoxib is taken orally at 200 mg per dose, twice daily, for a duration of 6 months.
Procedure: Curative resection of colorectal cancer — Patients who do not achieve cCR based on radiographic imaging (CT/MRI of chest, abdomen, pelvis, and rectal MRI), endoscopy, and digital rectal examination (if applicable) are recommended to undergo curative resection of colorectal cancer.
Other: Watch-and-wait strategy — Patients achieving clinical complete response (cCR) based on radiographic imaging (CT/MRI of chest, abdomen, pelvis, and rectal MRI), endoscopy, and digital rectal examination (if applicable) are recommended to adopt a watch-and-wait strategy.

SUMMARY:
Several Phase II studies have demonstrated the feasibility, effectiveness, and good tolerability of neoadjuvant immune checkpoint inhibitor (ICI) treatment for localized dMMR colorectal and rectal cancers. The significant clinical and pathological complete response rates offer the possibility of avoiding surgical resection. dMMR colorectal cancers are generally larger and more advanced than pMMR tumors, often requiring more extensive surgery with associated risks such as anastomotic leakage, ureteral injury, and infection. If oncological outcomes are not affected (requiring long-term follow-up), non-surgical treatment becomes an attractive option for localized dMMR colorectal cancer. Moreover, pelvic radiotherapy, the standard for locally advanced rectal cancer, causes both short-term and long-term adverse effects (e.g., bowel and bladder dysfunction, fistula, infertility), significantly impacting quality of life. Total mesorectal excision also carries risks of complications and sexual dysfunction, often requiring a stoma, making organ preservation a more urgent need for rectal cancer patients.

Phase II trials and the international "watch-and-wait" database have confirmed the feasibility and safety of organ preservation for pMMR locally advanced rectal cancer. Therefore, the high clinical and pathological complete response rates achieved by neoadjuvant immunotherapy for dMMR/MSI-H rectal cancer offer promising prospects for non-surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and willingness/compliance with study procedures.
2. Age ≥18 years.
3. Histologically confirmed colorectal adenocarcinoma.
4. ECOG performance status 0-1.
5. Locally advanced primary tumor (T3/T4 and/or N+) confirmed by CT/MRI (pelvic MRI for rectal cancer).
6. dMMR (IHC) or MSI-H (PCR) status.
7. No prior anti-cancer therapy for colonrectal cancer (surgery/chemotherapy/targeted therapy/radiation).
8. Adequate organ function
9. For women of childbearing potential: negative pregnancy test and contraception use during and for 3 months post-treatment. Male participants with fertile partners must use contraception.
10. Willingness to adhere to study requirements.

Exclusion Criteria:

1. Presence of distant metastases (M1) confirmed by CT/MRI or PET-CT (at least covering the chest, abdomen, and pelvis).
2. Complete intestinal obstruction, active bleeding, or perforation requiring emergency surgery.
3. Inability to achieve complete resection of the primary colorectal tumor.
4. History or concurrent active malignancy (except malignancies cured ≥5 years ago or adequately treated carcinoma in situ).
5. Prior treatment with anti-PD-1/PD-L1 antibodies, anti-CTLA-4 antibodies, or other drugs/antibodies targeting T-cell co-stimulation or checkpoint pathways.
6. Major surgery (e.g., laparotomy, thoracotomy, organ resection via laparoscopy) or severe trauma within 4 weeks before enrollment (surgical incision must be fully healed).
7. Thromboembolic events (e.g., cerebrovascular accident, transient ischemic attack, pulmonary embolism, deep vein thrombosis) within 12 months before enrollment.
8. Active coronary artery disease, severe/unstable angina, or newly diagnosed angina/myocardial infarction within 12 months before enrollment.
9. New York Heart Association (NYHA) Class II or higher congestive heart failure (see Appendix 3).
10. HIV infection, AIDS, or untreated active hepatitis (HBV-DNA ≥500 IU/mL; HCV-RNA above detection limit).
11. Active inflammatory bowel disease or other colorectal disorders causing chronic diarrhea.
12. Active, known, or suspected autoimmune disease (exceptions: stable conditions like type 1 diabetes, hypothyroidism on hormone replacement, or skin disorders without systemic treatment, e.g., vitiligo, psoriasis, alopecia).
13. Interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, acute pneumonia).
14. Residual toxicity ≥Grade 2 (per CTCAE v5.0) from prior therapies (except anemia, alopecia, skin pigmentation).
15. Known or suspected hypersensitivity to any study-related drugs.
16. Pregnancy or lactation.
17. Women of childbearing potential (last menstruation <2 years ago) or fertile men unwilling to use effective non-hormonal contraception.
18. Any unstable medical condition compromising safety or protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 3 years
  the time between randomization and one of the following events: locally progressive disease leading to an unresectable tumor, local R2 resection, local recurrence after an R0/1 resection, distant metastases, a new primary colorectal cancer, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) rate | 3 years
  the percentage of subjects with no residual viable tumor in the resected primary tumor specimen and all sampled regional lymph nodes after radical surgery (ypT0N0).
Overall survival (OS) | 3 years
  the time from randomization to death from any cause. Subjects who are still alive at the time of the analysis will be censored for OS on the latest known survival date.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No